CLINICAL TRIAL: NCT05561543
Title: Effects of Peppermint Oil in Cardiometabolic Outcomes in Participants With Mild-moderate Hypertension.
Brief Title: Effects of Peppermint Oil in Mild-moderate Hypertension.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Collaborators: University of Hertfordshire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Peppermint oil hypertension
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — peppermint oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Identical in taste and colour to the supplement juice, but with no peppermint content.
  Interventions: Other: Placebo
- Peppermint oil (Experimental): 50 uL of peppermint oil, which will be diluted with 100 mL of water - taken twice per day.
  Interventions: Dietary Supplement: Peppermint oil

INTERVENTIONS:
Dietary Supplement: Peppermint oil — Peppermint oil
  Arms: Peppermint oil
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Cardiovascular and associated hypertensive diseases are the leading health burden and cause of mortality worldwide; therefore, the necessity for effective interventions is paramount. Dietary interventions to improve cardiovascular health are highly sought after as they possess less risk and financial burden than pharmacological drugs. Our previous randomized trial has shown that oral peppermint can improving systolic blood pressure and other cardiovascular/ blood lipids in healthy individuals. However, to date, no research has explored this using a placebo randomized intervention in patients with hypertension.

Therefore, the primary purpose of the proposed investigation is to test the ability of oral peppermint oil supplementation to improve cardiometabolic parameters in participants with mild-moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18-65 years
2. Systolic blood pressure 120 to 139 mmHg
3. Not taking prescribed medicine for blood pressure management
4. have the ability to complete written questionnaires independently
5. Able to provide informed consent

Exclusion Criteria:

1. diagnosed diabetes mellitus
2. known cardiovascular disease or clinically significant cardiovascular comorbidity, including coronary heart disease, symptomatic heart failure, clinically significant arrhythmia, or a history of stroke or transient ischaemic attack within the previous 6 months
3. known or suspected secondary hypertension, including renal, renovascular, or endocrine causes
4. known clinically significant renal impairment or severe hepatic disease
5. evidence or history of severe hypertension related target organ damage requiring specialist management
6. pregnant or lactating women
7. allergy to peppermint
8. habitual consumption of peppermint products
9. regular consumption of antioxidant supplements
10. body mass index larger than 40.0 kg/m²
11. current enrolment in other clinical trials or use of other external therapies likely to influence outcomes
12. condition(s) likely to compromise informed consent, protocol compliance, or outcome assessment, including severe psychiatric illness, cognitive impairment, or active substance or alcohol misuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | Baseline
  Systolic blood pressure - measured using a digital blood pressure monitor
Systolic blood pressure | 20 days
  Systolic blood pressure - measured using a digital blood pressure monitor

SECONDARY OUTCOMES:
Diastolic blood pressure | Baseline
  Diastolic blood pressure - measured using a digital blood pressure monitor
Diastolic blood pressure | 20 days
  Diastolic blood pressure - measured using a digital blood pressure monitor
Percent bodyfat and fat mass | Baseline
  Participants percentage composition of fat - measured using bio-electrical impedance
Percent bodyfat and fat mass | 20 days
  Participants percentage composition of fat - measured using bio-electrical impedance
Waist circumference | Baseline
  Waist circumference - measured using anthropocentric tape
Waist circumference | 20 days
  Waist circumference - measured using anthropocentric tape
Waist to hip ratio | Baseline
  Ratio of waist to hip circumference - measured using anthropocentric tape
Waist to hip ratio | 20 days
  Ratio of waist to hip circumference - measured using anthropocentric tape
Blood glucose | Baseline
  Capillary blood glucose - mmol/L
Blood glucose | 20 days
  Capillary blood glucose - mmol/L
Blood triglycerides | Baseline
  Capillary blood triglycerides - mmol/L
Blood triglycerides | 20 days
  Capillary blood triglycerides - mmol/L
Blood cholesterol (Total, HDL & LDL) | Baseline
  Capillary blood cholesterol - mmol/L
Blood cholesterol (Total, HDL & LDL) | 20 days
  Capillary blood cholesterol - mmol/L
Total and HDL cholesterol ratio | Baseline
  Ratio of total cholesterol to HDL cholesterol
Total and HDL cholesterol ratio | 20 days
  Ratio of total cholesterol to HDL cholesterol
LDL and HDL cholesterol ratio | Baseline
  Ratio of LDL to HDL cholesterol
Total and HDL cholesterol ratio | 20 days
  Ratio of LDL to HDL cholesterol
Triglyceride glucose index | Baseline
  Log transformed measurement of the blood glucose and blood triglyceride measures outlined above.
Triglyceride glucose index | 20 days
  Log transformed measurement of the blood glucose and blood triglyceride measures outlined above.
Coop-Wonka chart | Baseline
  Psychological wellbeing - The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Coop-Wonka chart | 20 days
  Psychological wellbeing - The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Beck Depression Inventory | Baseline
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
Beck Depression Inventory | 20 days
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
State Trait Anxiety Inventory | Baseline
  Psychological wellbeing - the state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
State Trait Anxiety Inventory | 20 days
  Psychological wellbeing - the state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
Insomnia Severity Index | Baseline
  Sleep quality - The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Insomnia Severity Index | 20 days
  Sleep quality - The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Pittsburgh Sleep Quality Index | Baseline
  Sleep quality - The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Pittsburgh Sleep Quality Index | 20 days
  Sleep quality - The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Epworth Sleepiness Scale | Baseline
  Sleep quality - The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.
Epworth Sleepiness Scale | 20 days
  Sleep quality - The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Lancashire, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sinclair J, Du X, Shadwell G, Dillon S, Butters B, Bottoms L. Effects of peppermint (Mentha piperita L.) oil in cardiometabolic outcomes in participants with pre and stage 1 hypertension: Protocol for a placebo randomized controlled trial. PLoS One. 2025 May 7;20(5):e0321986. doi: 10.1371/journal.pone.0321986. eCollection 2025. PMID 40333716